CLINICAL TRIAL: NCT03471169
Title: Studies on the Individualized Prevention of Cerebrovascular Disease Using Study on Antithrombotic Therapy in Beijing
Brief Title: Individualized Antithrombotic Therapy for Patients With Ischemic Cerebrovascular Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Chinese PLA General Hospital (Other); Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: jinqiaowml
Record Dates: First submitted 2017-12-05; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2017-11

CONDITIONS: Cerebrovascular Disease
Keywords: antithrombotic therapy
MeSH Terms: conditions — Cerebrovascular Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desirable TEG (Experimental): Patients receiving antiplatelet medication and desirable thrombelastogram(TEG) test results.
  Interventions: Drug: Desirable TEG
- Undesirable TEG (Sham Comparator): Patients receiving antiplatelet medication and undesirable thrombelastogram(TEG) test results.
  Interventions: Drug: Undesirable TEG

INTERVENTIONS:
Drug: Desirable TEG — Change the type and dose of antithrombotic therapy and obtain desirable TEG results.
  Antithrombotic drugs inclued Bayaspirin®，Plavix ® and Cilostazol.
  Other Names: blood sampling
  Arms: Desirable TEG
Drug: Undesirable TEG — Don't change the type and dose of antithrombotic therapy and obtain undesirable TEG results. Antithrombotic drugs inclued Bayaspirin®，Plavix ® and Cilostazol.
  Other Names: blood sampling
  Arms: Undesirable TEG

SUMMARY:
To investigate the therapeutic effect of individualized treatment of antiplatelet in secondary prevention of ischemic stroke.

DETAILED DESCRIPTION:
Ischemic stroke is a leading cause of disability and death worldwide. Antiplatelet treatment is one of treatment strategies in secondary stroke prevention for patients with non-cardioemoblism etiology. However, a concerning issue is that wide interindividual variability in P2Y12 antagonist, especially clopidogrel. The rate on-treatment high platelet reactivity (HPR) can be as high as in one-third of patients with standard dose of clopidogrel( i.e. 75mg), and HPR has been noted in those who received other P2Y12 antagonists, such as ticagrelor and prasugrel. In the present study, we aimed to investigate the safety and potential therapeutic effect of individualized treatment of antiplatelet in secondary prevention in a cohort of patients with non-cardioembolic ischemic strokes.

ELIGIBILITY:
Inclusion Criteria:

* 14 years of age or older
* no gender aspirin or clopidogrel for ischemic cerebrovascular disease Primary or secondary prevention of ischemic stroke patients
* The researcher (or principal) signs the informed consent form

Exclusion Criteria:

* Significant head trauma or stroke in the last 3 months
* 3 months to accept intracranial, spinal surgery or other parts of large surgery
* In the last week there is an incurable part of the artery puncture
* Acute bleeding constitution, including platelet count <100 × 109 / L or other conditions
* within the last 48h heparin treatment, APTT higher than the upper limit of normal range
* Oral anticoagulant: INR> 1.7 or PT> 15s
* The presence of intracranial tumors, aneurysms or arteriovenous malformations
* Patients with any of the following cardioembolic-related illnesses are identified: rheumatic mitral or aortic stenosis, prosthetic heart valves, atrial fibrillation, atrial flutter, sick sinus syndrome, left atrial myxoma, Open foramen ovale, left ventricular mural thrombus or valvular vegetation, congestive heart failure, bacterial endocarditis, or any other cardiovascular disease not suitable for enrollment; (as determined by the investigator)
* Severe liver and kidney dysfunction
* Life expectancy is less than 1 year
* Pregnant or lactating women
* Participating in other clinical studies, or have participated in other clinical studies within the 3 months before enrolling, or have already participated in this research
* Allergic or intolerant to aspirin or clopidogrel
* There are stomach lesions, such as gastritis, gastric ulcer and so on
* Do not want to follow-up or poor treatment compliance

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficient Aspirin | one year
  The value of inhibition rate of Aspirin > 50%

SECONDARY OUTCOMES:
Efficient Clopidogrel | one year
  The value of adenosine diphosphate> 30%

OTHER OUTCOMES:
Platelet aggregability | one year
  The value of maximum extent of thrombosis around 31-47 mm

CONTACTS AND LOCATIONS:
Overall Officials: Qian Zhang, 1, Study Director — Xuanwu Hospital, Beijing
Locations (1):
- XuanWu hospital, Beijing, Xicheng, China

IPD SHARING:
Plan to Share IPD: No